CLINICAL TRIAL: NCT03176758
Title: Postoperative Pain in Total Knee Arthroplasty: a Comparison Between General and Spinal Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, David segal, Principle Investigator, Meir Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0094-17-MMC
Record Dates: First submitted 2017-05-21; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Total Knee Replacement Surgery
MeSH Terms: interventions — Anesthesia, Spinal; Anesthetics, General; Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: The participant will be non-randomly enrolled into two groups. The default treatment, which was found as the preferred method by numerous investigators will be offered to all participants. Those who will ask for the second option (general anesthesia) or those who will not be aligble for spinlal block will be enrolled in the second group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Spinal block (Active Comparator): Intrathecal 10 mg Heavy Marcaine, 200 mcg Morphine + High volume local anesthesia infiltration Bupivacaine 5mg/ml + adrenaline 5 mcg/ml 3mg/kg ideal body weight diluted with 100cc Normal Saline
  + Total Knee Replacement ( which will not be the intervention of interest)
  Interventions: Drug: Spinal Block; Device: Total knee replacement
- General anesthesia (Active Comparator): 1-3 mg IV propofol 0.5 mg/kg IV Rocuronium + Fentanyl 2-3 mcg/kg + Morphine 0.1mg/kg IV Maintenance: Volatile anesthetic + High volume local anesthesia infiltration Bupivacaine 5mg/ml + adrenaline 5 mcg/ml 3mg/kg ideal body weight diluted with 100cc Normal Saline
  + Total Knee Replacement ( which will not be the intervention of interest)
  Interventions: Drug: General anesthetic; Device: Total knee replacement

INTERVENTIONS:
Drug: Spinal Block — Intrathecal 10 mg Heavy Marcaine, 200 mcg Morphine + High volume local anesthesia infiltration Bupivacaine 5mg/ml + adrenaline 5 mcg/ml 3mg/kg IBW diluted with 100cc Normal Saline
  Other Names: Neurological block
  Arms: Spinal block
Drug: General anesthetic — 1-3 mg IV propofol 0.5 mg/kg IV Rocuronium + Fentanyl 2-3 mcg/kg + Morphine 0.1mg/kg IV Maintenance: Volatile anesthetic + High volume local anesthesia infiltration Bupivacaine 5mg/ml + adrenaline 5 mcg/ml 3mg/kg IBW diluted with 100cc Normal Saline
  Arms: General anesthesia
Device: Total knee replacement — A total knee arthroplasty surgery, which is not the intervention of interest

SUMMARY:
Total knee arthroplasty may be conducted either under general anesthesia or spinal block. previous studies have shown that spinal block leads to less complications. The investigators aim to find whether post-operative pain is also diminished under spinal block compared to general anesthesia

DETAILED DESCRIPTION:
Patients who will be registered for a total knee replacement in Meir Medical Center and that will agree to participate in the study will be enrolled into one of two groups: the first, which will be the default choice for all patients, will be operated under a spinal block. Patients who will ask specifically for general anesthesia, or those in which the anesthesiologist will prefer general anesthesia due to medical reasons will be enrolled into the second group. For both groups the surgeon will add intraoperative peri-articular infiltration of local Marcaine injections, which was previously shown to diminish postoperative pain. The postoperative pain will be evaluated with the Visual Analogue Scale at different point during the first 48 hours following operation. Physiotherapy achievements will also be recorded. The investigators will try to find whether one of the two groups suffered less pain or had achieved better results in physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* all patient who will undergo total knee arthroplasty

Exclusion Criteria:

* patients who will not agree to participate in the study
* patients who will die during the research timeframe

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain measured by Visual Analogue Scale | 48 hours
  Visual Analogue Scale scores of pain will be documented at different timed during the first 48 postoperative hours

SECONDARY OUTCOMES:
Achievements in physical therapy measured by walking distance on the first postoperative day | 24 hours
  The patient will walk with a walker under the surgeon's supervision, and the surgeon will measure with the distance the succeeded walking

IPD SHARING:
Plan to Share IPD: No
Participant's data will be collectively statistically analyzed, The results will be available as part of the researches findings while the participant's information will not be shared.

REFERENCES:
- [Background] Turnbull ZA, Sastow D, Giambrone GP, Tedore T. Anesthesia for the patient undergoing total knee replacement: current status and future prospects. Local Reg Anesth. 2017 Mar 8;10:1-7. doi: 10.2147/LRA.S101373. eCollection 2017. PMID 28331362
- [Background] Kwofie MK, Shastri UD, Gadsden JC, Sinha SK, Abrams JH, Xu D, Salviz EA. The effects of ultrasound-guided adductor canal block versus femoral nerve block on quadriceps strength and fall risk: a blinded, randomized trial of volunteers. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):321-5. doi: 10.1097/AAP.0b013e318295df80. PMID 23788068
- [Background] Manickam B, Perlas A, Duggan E, Brull R, Chan VW, Ramlogan R. Feasibility and efficacy of ultrasound-guided block of the saphenous nerve in the adductor canal. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):578-80. doi: 10.1097/aap.0b013e3181bfbf84. PMID 19916251
- [Background] Macfarlane AJ, Prasad GA, Chan VW, Brull R. Does regional anesthesia improve outcome after total knee arthroplasty? Clin Orthop Relat Res. 2009 Sep;467(9):2379-402. doi: 10.1007/s11999-008-0666-9. Epub 2009 Jan 7. PMID 19130163
- [Background] Busch CA, Shore BJ, Bhandari R, Ganapathy S, MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW. Efficacy of periarticular multimodal drug injection in total knee arthroplasty. A randomized trial. J Bone Joint Surg Am. 2006 May;88(5):959-63. doi: 10.2106/JBJS.E.00344. PMID 16651569
- [Background] Memtsoudis SG, Sun X, Chiu YL, Stundner O, Liu SS, Banerjee S, Mazumdar M, Sharrock NE. Perioperative comparative effectiveness of anesthetic technique in orthopedic patients. Anesthesiology. 2013 May;118(5):1046-58. doi: 10.1097/ALN.0b013e318286061d. PMID 23612126